CLINICAL TRIAL: NCT01692041
Title: Tolerance and Effect of an add-on Treatment With a Cough Medicine Containing Ivy Leaves Dry Extract on Lung Function in Children With Bronchial Asthma
Brief Title: Effect of an add-on Treatment With Ivy Leaves Dry Extract on Lung Function in Bronchial Asthma
Acronym: HeHe
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HeHe
Record Dates: First submitted 2012-05-03; First posted 2012-09-25 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Asthma
Keywords: asthma; children
MeSH Terms: conditions — Asthma | interventions — EA 575 extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivy leave (Active Comparator): active therapy arm with Ivy leave 5 ml twice daily p.o. for four weeks
  Interventions: Drug: ivy leaves dry extract
- Placebo (Placebo Comparator): Ivy leave placebo 5 ml twice daily p.o. for four weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ivy leaves dry extract — 5 ml twice daily po
  Arms: Ivy leave
Drug: Placebo — 5 ml per os twice daily
  Arms: Placebo

SUMMARY:
The trial aims to record possible effects of a supplementary treatment with ivy leaves dry extract on different lung function parameter, on bronchial hyperreactivity, on individual markers of asthmatic inflammation and on the clinical symptom profile. The hypothesis is, that the additional therapy might improve these parameters and might help to optimize asthma therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Medical diagnosis of uncontrolled, mild, persistent, allergic bronchial asthma in terms of the bronchial asthma NVL Version 1.3 (2011)
2. Children aged from 6 to 12 years (girls and boys)
3. Signed Informed Consent of the patient and his legal guardians to participate in the trial after written and verbal briefing by the Investigator
4. Improvement of the FEV1≥12% after 2 puffs of terbutaline 100 µg dur-ing steroid monotherapy with 400 µg budesonide equivalent/day or an ACT score ≤ 19 as an indication of insufficient asthma control
5. Asthma diagnosis for at least 1 year

Exclusion Criteria:

1. Anamnestically known intolerance/allergy to one of the drugs applied or to their ingredients or to drugs of similar chemical structure
2. Participation of the patient in another clinical trial within the last four weeks before enrollment in this trial
3. Evidence suggesting that the patient or their legal representative is not likely to follow the trial protocol (e.g. lacking compliance)
4. Inability to measure lung function, to test bronchospasmolysis, to determine FeNO or to collect exhaled breath condensate, inability to document the symptoms in a symptom log book or questionnaire; in-ability to take the trial medication properly
5. Chronic illnesses of different aetiology
6. Vocal cord dysfunction
7. Premature birth or diagnosis of bronchopulmonary dysplasia
8. Gastroesophageal reflux
9. Acute respiratory infection within the previous 4 weeks
10. Hereditary fructose intolerance
11. Pregnant or breastfeeding girls -

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
MEF75-25 before bronchodilation - relative change | every 4 weeks
  MEF75-25 will be measured at every time point of the study and relative changes will be followed
FEV1 before bronchodilation - relative change | every 4 weeks
  FEV1 before bronchodilation will be measured at every study visit and changes will be documented

SECONDARY OUTCOMES:
MEF75-25 before bronchodilation - absolute change | every 4 weeks
FEV1 before bronchodilation - absolute change | every 4 weeks
  FEV1 before bronchodilation will be measured every visit and changes documented
Emergency treatment (beta agonist demand) | daily
  Emergency treatment (beta agonist demand)will be documented daily at home and checked at every study visit
Number of days with asthma symptoms | daily
  Number of days with asthma symptoms will be documented daily and checked at every study visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Carl Gustav Carus, Kinderklinik, Dresden, Saxony, Germany